CLINICAL TRIAL: NCT01087918
Title: Effects of Automated Treadmill Training and Lower Extremity Strength Training on Walking-related and Other Outcomes in Subjects With Chronic Incomplete Spinal Cord Injury
Brief Title: Lokomat Versus Strength Training in Chronic Incomplete Spinal Cord Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: EK-21/2008; CLI006/2 extension (Other Grant/Funding Number: Spinal Research)
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Results first posted 2012-10-19 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Spinal Cord Injury
Keywords: ASIA C and D
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- First RAGT, then strength training (Experimental): 16 sessions of 45 minutes of robot-assisted gait training 4 times a week in first intervention period and 16 sessions of 45 minutes of strength training 4 times a week in second intervention period.
  Interventions: Device: RAGT; Other: Strength Training
- First strength training, then RAGT (Experimental): 16 sessions of 45 minutes of strength training 4 times a week in first intervention period and 16 sessions of 45 minutes of robot-assisted gait training 4 times a week in second intervention period.
  Interventions: Device: RAGT; Other: Strength Training

INTERVENTIONS:
Device: RAGT — 16 sessions / 4 times/week / 45 minutes Lokomat training
Other: Strength Training — 16 sessions / 4 times/week / 45 minutes lower extremity strength training

SUMMARY:
The purpose of this pilot study is to investigate whether gait specific robotic supported bodyweight supported treadmill training and lower extremity strength training have similar beneficial effects on walking function and other outcomes.

DETAILED DESCRIPTION:
Although task-specific training has been promoted during the last years to improve function, recent studies showed that after an incomplete spinal cord injury, strength, but not complex movement coordination, is affected. In this randomized cross-over trial we investigate the effectiveness of a task-specific 4 week Lokomat training with a 4 week (unspecific) lower extremity muscle strength training on walking-related and other outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Time since lesion > 1 year
* Outdoor mobility SCIM III < 5
* Stable walking capacity

Exclusion Criteria:

* participating on other training studies
* osteoporosis
* psychiatric diseases
* epilepsia
* body weight > 130 kg
* cardiac pacemaker

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huub van Hedel, PhD, Principal Investigator — University of Zurich
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Labruyere R, van Hedel HJ. Strength training versus robot-assisted gait training after incomplete spinal cord injury: a randomized pilot study in patients depending on walking assistance. J Neuroeng Rehabil. 2014 Jan 9;11:4. doi: 10.1186/1743-0003-11-4. PMID 24401143

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant recruitment from a spinal cord injury hospital in Zurich, Switzerland between March 2009 and March 2011.
Pre-assignment Details: 97 possible participants recruited; 9 participated, 88 excluded (12 did not meet inclusion criteria and 76 refused participation)
Groups:
- Robot-assisted Gait Training First, Then Strength Training: 16 sessions of 45 minutes of robot-assisted gait training 4 times a week in first intervention period and 16 sessions of 45 minutes of strength training 4 times a week in second intervention period.
- Strength Training First, Then Robot-assisted Gait Training: 16 sessions of 45 minutes of strength training 4 times a week in first intervention period and 16 sessions of 45 minutes of robot-assisted gait training 4 times a week in second intervention period.
Period: Overall Study
Arm/Group | Robot-assisted Gait Training First, Then Strength Training | Strength Training First, Then Robot-assisted Gait Training
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Robot-assisted Gait Training First, Then Strength Training | Strength Training First, Then Robot-assisted Gait Training | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 2 | 2 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 58.8 (11.1) | 59.3 (12.8) | 59.0 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  Switzerland | 4 | 3 | 7
  Germany | 1 | 1 | 2
Weight [Mean (Standard Deviation); unit: kg] | 80.8 (15.9) | 70.0 (17.1) | 76.0 (16.4)
Height [Mean (Standard Deviation); unit: m] | 1.76 (0.077) | 1.67 (0.075) | 1.72 (0.086)

OUTCOME MEASURES:

1. Primary Outcome: 10 Meter Walking at Preferred Speed
Description: The 10 meter walk test assesses the time required to walk 10 meters at the patient's preferred speed (in seconds). Results were converted to walking speed [m/s]. Displayed are values after each intervention (RAGT or strength training) minus value at baseline. Positive values denote improvements.
Time Frame: Baseline, after intervention (4 weeks)
Measure: Mean (Standard Deviation); unit: meters per second
Groups:
- Robot-assisted Gait Training; Strength Training: 16 sessions of 45 minutes of robot-assisted gait training 4 times a week.
Arm/Group | Robot-assisted Gait Training | Strength Training
Number analyzed (Participants) | 9 | 9
meters per second | 0.04 (0.10) | 0.06 (0.08)

2. Secondary Outcome: Walking Index for Spinal Cord Injury II
Description: The WISCI II describes whether a patients requires waling aids, braces or personal assistance to walk 10 meters. It is an ordinal scale varying from 0 (= not able to walk 10 meters) to 20 (= able to walk 10 meters with no walking aids, braces or personal assistance). Displayed are values after each intervention (RAGT or strength training) minus value at baseline. Positive values denote improvements.
Time Frame: Baseline, after intervention (4 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Robot-assisted Gait Training | Strength Training
Number analyzed (Participants) | 9 | 9
units on a scale | 0.78 (1.6) | 0.33 (1.0)

3. Secondary Outcome: Berg Balance Scale
Description: The Berg Balance Scale is a performance-based measure of balance. It is scored from 0 (= failed all items) to 56 points (= scored maximally in all items). Displayed are values after each intervention (RAGT or strength training) minus value at baseline. Positive values denote improvements.
Time Frame: Baseline, after intervention (4 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Strength Training: 16 sessions of 45 minutes of strength training 4 times a week
Arm/Group | Robot-assisted Gait Training | Strength Training
Number analyzed (Participants) | 9 | 9
units on a scale | 1.11 (1.90) | 2.78 (1.92)

4. Secondary Outcome: Spinal Cord Independence Measure III
Description: The SCIM assesses functional independence after spinal cord injury. It is scored from 0 (= total dependence in everyday life) to 100 points (= complete independence in everyday life). Displayed are values after each intervention (RAGT or strength training) minus value at baseline. Positive values denote improvements.
Time Frame: Baseline, after intervention (4 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Robot-assisted Gait Training | Strength Training
Number analyzed (Participants) | 9 | 9
units on a scale | 0.78 (2.17) | 1.33 (1.87)

5. Secondary Outcome: Mean Latency of the Averaged Motor Evoked Potentials of the Right and the Left M. Tibialis
Description: Motor evoked potential was elicited by transcranial magnetic stimulation. Displayed are values after each intervention (RAGT or strength training) minus value at baseline. Negative values denote improvements.
Time Frame: Baseline, after intervention (4 weeks)
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Robot-assisted Gait Training | Strength Training
Number analyzed (Participants) | 9 | 9
milliseconds | 0.43 (1.42) | 0.42 (1.38)

6. Secondary Outcome: Manual Muscle Test of the Lower Extremity
Description: With the manual muscle test, we examined strength of the lower extremities. Five key muscles on each side are evaluated from 0 (= total paralysis) to 5 (= normal strength). Values for left and right were then averaged. Displayed are values after each intervention (RAGT or strength training) minus value at baseline. Positive values denote improvements.
Time Frame: Baseline, after intervention (4 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Robot-assisted Gait Training | Strength Training
Number analyzed (Participants) | 9 | 9
units on a scale | 0.67 (1.12) | 1.00 (1.00)

7. Secondary Outcome: Pain on a Visual Analogue Scale
Description: Pain was scored on a visual analogue scale from 0 (= no pain) to 100 (= maximal pain). Displayed are values after each intervention (RAGT or strength training) minus value at baseline. Negative values denote improvements.
Time Frame: Baseline, after intervention (4 weeks)
Population: Only 8 patients participated at pain assessments as 1 patient did not suffer from pain.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Robot-assisted Gait Training | Strength Training
Number analyzed (Participants) | 8 | 8
units on a scale | -4.5 (2.2) | -6.8 (2.5)

8. Secondary Outcome: Response Time of the Lower Extremities
Description: We measured choice stepping response time on a plate in a standing position. Participant had to move their feet to flashing LEDs as fast as possible. Valid values of the right and the left foot were averaged. Displayed are values after each intervention (RAGT or strength training) minus value at baseline. Negative values denote improvements.
Time Frame: Baseline, after intervention (4 weeks)
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Robot-assisted Gait Training | Strength Training
Number analyzed (Participants) | 9 | 9
milliseconds | -1.8 (63.0) | -17.6 (66.4)

9. Secondary Outcome: Falls Efficacy Scale
Description: The Falls Efficacy Scale evaluates fear of falling in everyday life situations. It is scored from 16 (= no fear at all) to 64 points (= maximal fear in all items). Displayed are values after each intervention (RAGT or strength training) minus value at baseline. Negative values denote improvements.
Time Frame: Baseline, after intervention (4 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Robot-assisted Gait Training | Strength Training
Number analyzed (Participants) | 9 | 9
units on a scale | 0.17 (4.99) | 0.56 (2.88)

10. Primary Outcome: 10 Meter Walking at Maximal Speed
Description: The 10 meter walking speed assesses the time needed to walk 10 meters at maximal speed (in seconds). Results were converted to walking speed [m/s]. Displayed are values after each intervention (RAGT or strength training) minus value at baseline. Positive values denote improvements.
Time Frame: Baseline, after intervention (4 weeks)
Measure: Mean (Standard Deviation); unit: meters per second
Groups:
- First RAGT, Then Strength Training; First Strength Training, Then RAGT: 16 sessions of 45 minutes of robot-assisted gait training 4 times a week.
Arm/Group | First RAGT, Then Strength Training | First Strength Training, Then RAGT
Number analyzed (Participants) | 9 | 9
meters per second | 0.01 (0.18) | 0.14 (0.12)

11. Secondary Outcome: Figure of Eight Test
Description: The Figure of Eight Test is a 10m Walk Test in the shape of a figure of eight. Time for completion of one lap is recorded and converted to [m/s]. Displayed are values after each intervention (RAGT or strength training) minus value at baseline. Positive values denote improvements.
Time Frame: Baseline, after intervention (4 weeks)
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Robot-assisted Gait Training | Strength Training
Number analyzed (Participants) | 9 | 9
meters per second | 0.004 (0.04) | 0.04 (0.09)

ADVERSE EVENTS:
Arm/Group | Robot-assisted Gait Training First, Then Strength Training | Strength Training First, Then Robot-assisted Gait Training
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4

LIMITATIONS AND CAVEATS:
Issues to find participants led to small numbers of subjects analyzed. Ambulatory activity besides our interventions was not controlled for.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes